CLINICAL TRIAL: NCT04437979
Title: Association of Epicardial Fat Thickness and Inflammation With the Presence of Metabolic Syndrome in People With Obesity
Brief Title: Epicardial Fat Thickness and Inflammation in People With Metabolic Syndrome and Obesity
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Duygu Ersan Demirci, Principal investigator, Antalya Training and Research Hospital
Other Study IDs: 2019-397
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Metabolic Syndrome; Obesity; Inflammation
Keywords: epicardial fat thickness; metabolic syndrome; obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epicardial adipose tissue (EAT) is a type of visceral adipose tissue (VAT), functioning as a metabolically active endocrine organ and suggested to play an important role in the progression of metabolic syndrome (MetS). Obesity and MetS are commonly associated with an inflammatory status. The aim of the study was to evaluate the association of echocardiographically measured epicardial fat thickness (EFT) and inflammation, on the basis of c-reactive protein (CRP) and neutrophil-lymphocyte ratio (NLR), with MetS and its components in people with obesity.

A total of 104 patients with body mass index (BMI)≥30 kg/m² were enrolled to the study. In all participants, EFT was measured with transthoracic echocardiography at end-systole. The patients were then classified into two groups according to whether they had MetS or not. EFT, clinical and biochemical parameters were compared between the two groups

DETAILED DESCRIPTION:
Epicardial adipose tissue (EAT) is a kind of VAT, between the surface of the myocardium and the epicardium. It can easily be measured by standard two-dimensional (2D) echocardiography. EAT serves as an endocrin organ that secretes hormones, inflammatory cytokines and chemokines. Previous data suggests that EAT can play an active role in the development of metabolic syndrome (MetS). Previous studies have investigated the relationship between EAT/inflammatory markers and MetS/MetS components. However, there was lack of enough evidence regarding this relationship in people with obesity with or without MetS. The aim of the present study was to evaluate the association of echocardiographically measured EAT and inflammation, on the basis of c-reactive protein (CRP) and neutrophil-lymphocyte ratio (NLR), as simple and reliable indicators of inflammation, with MetS and its components in people with obesity who have similar body mass index (BMI) values. In this cross-sectional study, 104 consecutive patients with BMI ≥30 kg/m2 who presented to the 'Obesity Solution Center 'of Antalya Research and Training Hospital were included . Patients with manifest heart disease such as, coronary heart disease, cardiac failure, cardiac valve disease or arrythmia, renal failure, hepatic failure, infection, chronic systemic inflammatory disease, pulmonary disease , malignancy and inadequate transthoracic echocardiographic images were excluded. The study protocol was approved by the local ethics committee and informed consent was obtained from each subject.

Clinical information and current cardiovascular medication use were provided from each patient. Height, weight, waist circumference and hip circumference (HC) were measured when fasting and standing up with standard measuring tools. Patients were defined as having hypertension (HT) if their systolic blood pressure was >140 mmHg, their diastolic blood pressure was >90 mmHg, or they were using an antihypertensive medication. Blood samples were obtained after overnight fasting. Fasting blood glucose, urea, creatinine, total cholesterol, low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, triglycerides, CRP, fasting and postprandial insulin, C-peptid levels, vitamin D, ferritin and complete blood counts were measured using standard methods. Homeostasis model assessment of insulin resistance (HOMA-IR) was calculated using the method described by Matthews et al. NLR was defined as the log e neutrophil count/log e lymphocyte count within the peripheral blood. Patients were defined as having diabetes mellitus (DM) if they had a history of taking an oral antidiabetic or insulin medication, or if their fasting plasma glucose was ≥ 126 mg/dl. The patients were classified into two groups according to whether they had MetS or not. MetS was diagnosed according to the National Cholesterol Education Programme Adult Treatment Panel III (NCEP ATP III). Epicardial fat thickness (EFT) was identified as the echo-free space in the pericardial layers on 2D echocardiography. EFT was measured on the free wall of the right ventricle at end-systole from both parasternal long axis and parasternal short axis views using the mean of three consecutive beats.

ELIGIBILITY:
Inclusion Criteria:

- Having body mass index ≥30 kg/m2

Exclusion Criteria:.

* Manifest heart disease ( coronary heart disease, cardiac failure, cardiac valve disease or arrythmia)
* Renal failure
* Hepatic failure
* Infection
* Chronic systemic inflammatory disease
* Pulmonary disease
* Malignancy
* Inadequate transthoracic echocardiographic images

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with BMI ≥30 kg/m2, >18 years old and without manifest heart disease such as, coronary heart disease, cardiac failure, cardiac valve disease or arrythmia, renal failure, hepatic failure, infection, chronic systemic inflammatory disease, pulmonary disease and malignancy
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Estimation of the epicardial fat thickness in the presence of metabolic syndrome in people with obesity | 1 week
  Transthoracic echocardiography was performed to all participants with body mass index > 30 kg/m2 and epicardial fat thickness was measured. Epicardial fat thickness (EFT) was identified as the echo-free space in the pericardial layers on 2D echocardiography. EFT was measured on the free wall of the right ventricle at end-systole from both parasternal long axis and parasternal short axis views using the mean of three consecutive beats The patients were classified into two groups according to whether they had MetS or not. MetS was diagnosed according to the National Cholesterol Education Programme Adult Treatment Panel III. We evaluated the difference in epicardial fat thickness according to whether having metabolic syndrome or not, regardless of body mass index.

SECONDARY OUTCOMES:
Estimation of inflammation in the presence of metabolic syndrome in people with obesity | 1 week
  C-reactive protein and neutrophil-to-lymphocyte ratio were used to determine inflammation. The patients were classified into two groups according to whether they had MetS or not. MetS was diagnosed according to the National Cholesterol Education Programme Adult Treatment Panel III. We evaluated the difference in inflammatory mediators according to whether having metabolic syndrome or not, regardless of body mass index.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Ersan Demirci, MD, Principal Investigator — Antalya Research and Training Hospital
Locations (1):
- Antalya Research and Training Hospital, Antalya, Turkey (Türkiye)